CLINICAL TRIAL: NCT07335991
Title: Effect of Vitamin A Supplementation on the Onset and Progression of Idiopathic Scoliosis: A Prospective, Single-Blind, Randomized Controlled Trial
Brief Title: Effect of Vitamin A Supplementation on Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangyang Wang, M.D., Chief physician, Doctorial superviso, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2025-K-140-01
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Vitamin A Deficiency; Idiopathic Scoliosis
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiologists measuring Cobb angles will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin A Supplementation plus Nutritional Education (Experimental): 1. Dietary Supplement: A daily oral dose of 2000 IU Vitamin A (as retinyl palmitate or acetate) for 6 consecutive months.
  2. Behavioral: Nutritional Education: A one-time, standardized educational session at baseline delivered by a study dietitian. The session covers principles of a balanced diet for bone health, with a focus on food sources rich in vitamin A.
  Interventions: Dietary Supplement: Vitamin A
- Nutritional Education Only (Active Comparator): 1. Behavioral: Nutritional Education: An identical one-time, standardized educational session and materials as provided to Arm 1.
  2. No study-provided vitamin A supplements will be administered.
  Interventions: Behavioral: Nutritional Education

INTERVENTIONS:
Dietary Supplement: Vitamin A — Vitamin A supplements plus Nutritional Education
  Arms: Vitamin A Supplementation plus Nutritional Education
Behavioral: Nutritional Education — Nutritional Education Only
  Arms: Nutritional Education Only

SUMMARY:
This study aims to investigate whether vitamin A supplementation can influence spinal curve magnitude in idiopathic scoliosis children and potentially prevent its de novo development.

DETAILED DESCRIPTION:
Idiopathic scoliosis (IS) is the most common structural spinal deformity in children and adolescents. Despite extensive research, its etiology remains largely unknown, resulting in a lack of modifiable targets for prevention or early intervention. Notably, preliminary unpublished data from our pediatric health center indicate a high prevalence (up to 30%) of mild scoliosis among children with vitamin A deficiency. Furthermore, our pilot data suggest a tendency toward vitamin A insufficiency in many children diagnosed with IS. Vitamin A is critical for normal bone growth, embryonic skeletal development, and the maintenance of epithelial tissues. We hypothesize that chronic vitamin A deficiency may represent a modifiable risk factor that contributes to the pathogenesis or progression of IS by disrupting these fundamental processes.

This study will be conducted at the "Child Health-Spine Wellness" Center. Children with idiopathic scoliosis and concurrent vitamin A deficiency or insufficiency will be randomized into one of two groups. The Intervention Group will receive sustained biochemical correction through daily oral vitamin A supplementation (2000 IU) for 6 months, coupled with a standardized nutritional education session. The Control Group will receive an identical nutritional education session but no study-provided supplements, serving as an active comparator that controls for the effects of increased health awareness and general dietary advice. For all children with scoliosis, routine follow-up visits with radiographic assessment will be scheduled at 6-month intervals for at least 24 months to evaluate curve progression. Additionally, children with vitamin A deficiency but without scoliosis at baseline will also be randomized to the same supplementation regimens and will undergo annual scoliosis screening as part of an ongoing provincial health initiative. All participants will undergo serial radiographic and clinical assessments.

At the same time, a structured safety monitoring plan will be implemented to prevent and promptly identify both vitamin A deficiency persistence and hypervitaminosis A. Prior to randomization, all caregivers will receive standardized education on the signs and symptoms of both significant vitamin A deficiency (e.g., night blindness, dry eyes) and acute/chronic hypervitaminosis A (e.g., headache, nausea/vomiting, dizziness, blurred vision, skin dryness/peeling). They will be instructed to report any such symptoms immediately to the study team via a dedicated 24-hour contact line. Serum retinol concentration will be measured for all participants at baseline and the 6-month visit. This serves the dual purpose of monitoring adherence in the Long-term. If a participant's serum retinol level exceeds 1.0 mg/L, the study supplementation will be immediately suspended, and the participant will be referred to a pediatric nutritionist for further evaluation and management.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 15 years.
2. Biochemically confirmed vitamin A deficiency (serum retinol < 0.20 mg/L) or insufficiency (serum retinol 0.20-0.29 mg/L).
3. Has undergone radiographic evaluation (standing full-spine X-ray) for idiopathic scoliosis at the initial clinic visit.
4. Skeletally immature (Risser sign 0-3) with a major Cobb angle < 40 degrees at baseline.
5. Written informed consent/assent provided by the participant and legal guardian.

Exclusion Criteria:

1. Unwillingness or inability to comply with all study procedures and follow-up visits.
2. Plans to relocate outside the study area within the next 24 months.
3. Previous high-dose vitamin A supplementation therapy within the past 12 months.
4. Clinical signs of severe vitamin A deficiency syndrome (e.g., xerophthalmia, Bitot's spots).
5. Serum vitamin A level > 0.70 mg/L (to avoid risk of hypervitaminosis A).
6. Severe chronic health conditions that could confound study outcomes, including but not limited to:

   * Known syndromic, neuromuscular, or congenital musculoskeletal causes of scoliosis.
   * History of spine surgery or significant spinal trauma.
   * Spinal tumor.
   * Leg length discrepancy > 20 mm.
   * Other severe chronic diseases (e.g., poorly controlled diabetes, chronic liver or renal disease, malabsorption syndromes).
   * Severe obesity (body mass index z-score ≥ 3).

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Curve Angle | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  A long standard standing whole spine radiograph will be used for measuring curve size in terms of Cobb angle according to the standard Cobb method
Angle of Trunk Rotation | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  In addition to spinal X-rays, a Scoliometer can also help monitor curve progression. The Scoliometer is an inclinometer that measures the asymmetries between the sides of the trunk by measuring axial rotation in degrees. Numerous studies have found a high correlation between trunk axial rotation (ATR) values and the Cobb angles.

SECONDARY OUTCOMES:
Scoliosis Research Society-22 (SRS-22) questionnaire | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  The SRS-22 aims to evaluate health-related quality of life (HRQOL) in patients with idiopathic scoliosis. The SRS-22 specifically addresses areas affected by spinal deformities-such as pain, self-perception, function, mental health, and satisfaction with treatment. Consequently, it offers a focused approach to understanding the patient experience.
Change in Serum Vitamin A (Retinol) Level | At baseline and months 6
  Change in serum concentration of retinol (mg/L) measured by high-performance liquid chromatography (HPLC) between baseline and the 6-month visit.
Serum Levels of Vitamin D | At baseline and months 6
  Change in serum concentrations of Vitamin D potentially interacting with vitamin A metabolism or bone health from baseline to 6 months.
Change in Gene Expression Levels of biomarkers | At baseline and months 6
  Change in mRNA expression levels of specific Genes such as HIF1A, Bmal1 and IGFBPs in peripheral blood mononuclear cells (PBMCs) as measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR).
Circadian rhythm Measurements | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  Circadian rhythm as assessed by Morning and Evening Questionnaire-5 (MEQ-5)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided